CLINICAL TRIAL: NCT02970266
Title: Genetic Decryption of Leber Congenital Amaurosis (LCA) in a Large Cohort of Independent Families: Establishment of Genotype-phenotype Correlations and Updating the Clinical Definition of This Retinal Dystrophy
Brief Title: Genetic Decryption of Leber Congenital Amaurosis (LCA) in a Large Cohort of Independent Families.
Acronym: GENPHENACL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081257
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Leber Congenital Amaurosis
Keywords: Leber Congenital Amaurosis; Genetic Decryption; The genotype-phenotype correlations; Ethnicity families
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objectives of this study are:

1. Improve genetic counseling by establishment of prevalences of each of genetic subtypes within a expanded population of patients with LCA taking into account ethnicity of families.
2. Confirm, refine or modify the genotype-phenotype correlations.
3. Edit important recommendations for:

   * The clinical and paraclinical exploration of a new patient based on genotype, especially for extraocular explorations, to book at certain genetic subtypes
   * Prenatal care of a couple.
   * Directing families to a therapeutic protocol in progress or in development.
4. Individualize a panel of families without a mutation in the known genes and identify new genes responsible.

DETAILED DESCRIPTION:
This study characterize the clinical history of the disease (age and start mode of visual disturbances, rate and mode of progress of disease), careful assessment of retina function and finally, in search of the mutations responsible for this condition.

A full ophthalmic check-up, one at the inclusion and 24 months :

1. - A genetic consultation taking account of family history and establishment of family tree with precision of geographical origin of birth of ascendants.
2. - A thorough ophthalmologic examination by a referring medical ophthalmologist, including:

   2.1 - An interrogation on the development of the visual awakening since the birth and its possible disturbances.

   2.2 - The search for abnormal movements of the eyeballs, and difficulties with regard to different lighting.

   2.3 - Visual field evaluation Survey.

   2.4 - The study of color vision.

   2.5 - The search for a refractive disorder with the automatic refractometer.

   2.6 - Measurement of Visual acuity for near and distance.

   2.7 - Examination of the eyeball as a whole, examination of the anterior chamber of the eye by the slit lamp.

   2.8 - Taking pictures of the fundus of the eye after pupillary dilation.

   2.9 - An autofluorescence search using a Scanning Laser Ophthalmoscopy (SLO).

   2.10 - Optical Coherence Tomography (OCT) which used to assess the thickness of each of retinal layers.

   2.11 - Electrophysiological examination, Electroretinogram (ERG) that allows to record the functional value of the retina.

   These two latter examinations last on average 10 minutes after dilation of the pupil.
3. - A blood sample of 10 milliliters to carry out genetic studies to identify the gene responsible for this condition and genetic counseling refined by taking account the results of this study.

Intermediate visit M12: only for patients younger than 6 years of age on inclusion.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients of all ages
* Patients with symptoms the day of the first consultation allowing to ask the diagnosis of leber congenital amaurosis.
* Are affiliated to a social health care.
* Written informed consent must be given by patients or holders parental authority for minors.

patients and siblings:

* Signed consent for molecular study by the participant or by holders parental authority for minors.
* Are affiliated to a social health care.

Exclusion Criteria:

* Patients whose exploration has laid differential diagnoses.
* Patients refusing the visits provided for in Protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Leber Congenital Amaurosis (LCA) taking into account Ethnicity of families.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Improve genetic counseling by establishment of prevalences of each of genetic subtypes within a expanded population of patients with LCA. | 24 MONTHS

SECONDARY OUTCOMES:
Measurement of visual acuity using the logarithmic scale for children under 5 | 24 MONTHS
Measurement of visual acuity using Early Treatment Diabetic Retinopathy Study scale (ETDRS) for far vision | 24 MONTHS
The "Parinaud Scale" for near vision (After the age of 6) | 24 MONTHS
Visual field evaluation Survey | 24 MONTHS
Measurement of refraction by portable automatic refractometer. | 24 MONTHS
Screening for color vision abnormalities using "children's boards" of "Ishihara Test" from the age of 3-4. | 24 MONTHS
Screening for color vision abnormalities using "regular boards" as soon as learning to read figures from the age of five. | 24 MONTHS
Test the color vision deficiency using the " Farnsworth test" in adults and children after the age of 6. | 24 MONTHS
The visual field test using the Goldman dome in adults and children aged 6 to 7. | 24 MONTHS
Electrophysiological examination using Electroretinogram. | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Josseline KAPLAN, MD, Principal Investigator — Necker-Enfants Malades Hospital, 75015 Paris. France
Locations (1):
- Necker-Enfants Malades Hospital, Paris, Paris, France